CLINICAL TRIAL: NCT02668627
Title: MR-based Collateral Imaging to Predict Response to Endovascular Treatment of Stroke (FAST-COLL Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Oh Young Bang, Professor, Samsung Medical Center
Other Study IDs: SMC 2013-12-088
Record Dates: First submitted 2016-01-21; First posted 2016-01-29 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Stroke
Keywords: Stroke; Collateral status; Endovascular treatment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Endovascular treatment — Endovascular mechanical thrombectomy or endovascular delivery of thrombolytic agent

SUMMARY:
Based on the results of recent randomized controlled trials, current international guidelines recommend the initiation of endovascular treatment within 6 hours of symptom onset for acute ischemic stroke. Endovascular treatment may be beneficial in selected patients beyond 6 hour time window. In particular, treatment response to endovascular therapy may be greatly influenced by pretreatment collateral status. The aim of this study is to evaluate whether MRI-based collateral imaging (the Fast Analysis SysTem for COLLaterals, 'FAST-COLL') is feasible and can predict the response to endovascular treatment in a wide range of patients with acute ischemic stroke .

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke
* Age 20 years and older
* Disabling stroke defined as a baseline NIHSS > 5 at the time of arrival
* Onset (last-seen-well) time to endovascular treatment time < 12 hours
* Confirmed symptomatic intracranial occlusion, based on CT or MR angiography, at one or more of the following locations: Carotid T/L, M1 MCA, or M1-MCA equivalent (2 or more M2-MCAs)
* Signed informed consent or appropriate signed deferral of consent where approved

Exclusion Criteria:

* Baseline non-contrast CT reveals a moderate/large core defined as extensive early ischemic changes of ASPECTS 0-5 in the territory of symptomatic intracranial occlusion.
* Clinical history, past imaging or clinical judgment suggests that the intracranial occlusion is chronic
* Unable to undergo MRI (contraindicated or poor cooperation)
* Patient has a severe or fatal comorbid illness that will prevent improvement or follow-up or that will render the procedure unlikely to benefit the patient
* Pregnant females as determined by positive urine hCG test or lactating females

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke, eligible for endovascular treatment within 12 hours of symptom onset
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
90-days functional outcome | 90-days
  90-days modified Rankin Scale ≤ 2

SECONDARY OUTCOMES:
Early neurologic improvement | 24 hours
  An 8-point or more improvement on the NIH score when comparing the baseline score or a NIHSS score of 0-1, at 24 hours.
Symptomatic hemorrhagic transformation | During initial admission
  Occurrence of an increase in the National Institutes of Health Stroke Scale (NIHSS) score of 4 or more points in the setting of local or remote parenchymal hematoma.
Successful recanalization | within 24 hours of symptom onset
  Defined as modified Thrombolysis in Cerebral Infarction (mTICI) ≥ 2b

CONTACTS AND LOCATIONS:
Overall Officials: Oh Young Bang, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Yu I, Bang OY, Chung JW, Kim YC, Choi EH, Seo WK, Kim GM, Menon BK, Demchuk AM, Goyal M, Hill MD. Admission Diffusion-Weighted Imaging Lesion Volume in Patients With Large Vessel Occlusion Stroke and Alberta Stroke Program Early CT Score of >/=6 Points: Serial Computed Tomography-Magnetic Resonance Imaging Collateral Measurements. Stroke. 2019 Nov;50(11):3115-3120. doi: 10.1161/STROKEAHA.119.026229. Epub 2019 Sep 26. PMID 31554502